CLINICAL TRIAL: NCT06269835
Title: Intermittent Multifunctional Nutrition Tube Versus Persistent Nasogastric Tube Feeding in Infants With Cerebral Palsy and Dysphagia: A Randomized Controlled Study
Brief Title: Intermittent Multifunctional Nutrition Tube in Cerebral Palsy and Dysphagia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Head of R&D, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NAOTAN-IOE
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The observation group (Experimental): All participants were given routine rehabilitation treatment by professional rehabilitation therapists, including exercise therapy, guided education, psychological therapy, acupuncture and massage therapy, to promote the development of motor and cognitive function, as well as to improve intellectual development. Besides, swallowing function training was also provided, including direct training, indirect training, and compensatory training.Within 4 hours of admission, the observation group were required to undergo nasogastric tube removal and initiated Intermittent Oro-Esophageal Tube Feeding for nutrition support.
  Interventions: Behavioral: systemic therapy; Device: Intermittent Oro-Esophageal Tube Feeding
- The control group (Active Comparator): All participants were given routine rehabilitation treatment by professional rehabilitation therapists, including exercise therapy, guided education, psychological therapy, acupuncture and massage therapy, to promote the development of motor and cognitive function, as well as to improve intellectual development. Besides, swallowing function training was also provided, including direct training, indirect training, and compensatory training.The control group was given nutrition support with persistent nasogastric tube feeding , of which the tube passed through the nasal cavity into the stomach.
  Interventions: Behavioral: systemic therapy; Device: Persistent Nasogastric Tube Feeding

INTERVENTIONS:
Behavioral: systemic therapy — All participants were given routine rehabilitation treatment by professional rehabilitation therapists, including exercise therapy, guided education, psychological therapy, acupuncture and massage therapy, to promote the development of motor and cognitive function, as well as to improve intellectual development[. Besides, swallowing function training was also provided, including direct training, indirect training, and compensatory training, as follows The mendelson maneuver: performed 5 days per week, twice per day, 5-10 minutes each time.
  Cold stimulation of the pharynx: performed every day, twice per day, 3-5 minutes each time.
  Passive head extension: to stretch the submental muscle for 2-3 seconds, with upward resistance applied to the lower cheek for no less than 5 times a day and no less than 5 minutes each time.
  Direct feeding training: with powdered milk, once a day, 5 days a week.
Device: Intermittent Oro-Esophageal Tube Feeding — Within 4 hours of admission, the observation group were required to undergo nasogastric tube removal and initiated Intermittent Oro-Esophageal Tube Feeding for nutrition support. Before each feeding, the infant should rest for approximately 1 hour and undergo oral clean. During feeding, the infant should be held by the caregiver in a semi-reclined or upright position. Firstly, the tail of the tube was inserted via mouth into the upper part of the esophagus with a depth of 18-20cm, and the external part of the tube should be placed in water with the absence of bubbles indicating the successful tube placement. Subsequently, 1ml of water was slowly injected, followed by liquid food or water at a rate of approximately 50ml/min through a syringe connected to the feeding tube. After feeding, the tube should be slowly removed, and the feeding position should be maintained for 30-60 minutes to prevent reflux.
  Arms: The observation group
Device: Persistent Nasogastric Tube Feeding — The control group was given nutrition support with Persistent Nasogastric Tube Feeding, of which the tube passed through the nasal cavity into the stomach. After successful intubation, the tube was secured on the cheek. Liquid food was then syringe-fed into the stomach and the feeding was conducted every 2-3 hours, with each meal not exceeding 200 ml. The daily intake was generally consistent with that of the observation group. Besides, after successful intubation, the tube was secured on the infant's face and changed every one to two weeks.
  Arms: The control group

SUMMARY:
This was a randomized controlled study including 80 infants with cerebral palsy and dysphagia. The Participants were evenly divided into the observation group (with intermittent oro-esophageal tube feeding, n=40) and the control group (with persistent nasogastric tube feeding , n=40). Nutritional status and physical development, condition of dysphagia, and pneumonia before and after 3-month treatment were compared.

DETAILED DESCRIPTION:
In China, for nutrition support in the infants under one year of age with cerebral palsy and dysphagia, persistent nasogastric tube feeding is the mainstream choice. However, the efficacy of persistent nasogastric tube feeding is not sufficiently satisfactory, necessitating the exploration for a more effective and safe nutrition support approach. Therefore, this study reports the clinical effect of intermittent oro-esophageal tube feeding compared to persistent nasogastric tube feeding in the infants with cerebral palsy and dysphagia who received systemic therapy.

Method This was a randomized controlled study including 80 infants with cerebral palsy and dysphagia. The Participants were evenly divided into the observation group (with intermittent oro-esophageal tube feeding, n=40) and the control group (with persistent nasogastric tube feeding, n=40). Nutritional status and physical development, condition of dysphagia, and pneumonia before and after 3-month treatment were compared.

ELIGIBILITY:
Inclusion Criteria:

* meeting the diagnostic criteria of cerebral palsy formulated by the 13th National Conference on Pediatric Cerebral Palsy Rehabilitation;
* age<1 year;
* diagnosed as dysphagia confirmed by Dysphagia Disorder Survey or pediatric esophagoscopy;
* with a nasogastric tube inserted at admission;
* enteral nutrition support is required and feasible.

Exclusion Criteria:

* with dysphagia caused by other diseases or factors;
* with progressive neurological disease or degenerative neurological disease;
* with severe heart disease, liver or kidney dysfunction, hematological disorders, or other acute and severe symptoms;
* with abnormalities in the oral cavity, pharynx, esophagus, or other parts of the digestive tract;
* with poor compliance.

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The Oral Motor Assessment Scale | day 1 and day 90
  The Oral Motor Assessment Scale was a reliable and accurate scale. It consists of seven items compromising oral-motor skills. The assessment was conducted with the child in comfortable supported sitting with the head neutral position. The caregiver was allowed to feed the child one of the following foods normally: fed with a spoon soft food as yoghurt, a solid food as cookie or fed a liquid food with a glass, with/without a straw. The assessment primarily focused on feeding with 5 types of food (mash, semi-solids, solids, cracker, and liquid bottle/cup). Throughout the assessment, the examiner didn't interfere with the way the caregiver fed the child but just observed and scored each item of feeding process including chewing, sucking and swallowing. Each item of The Oral Motor Assessment Scale takes 30 second to be scored as passive (0), sub-functional (1), semi-functional (2) and functional (3). The final score was positively proportional to swallowing function.

SECONDARY OUTCOMES:
Pneumonia | day 1 and day 90
  The number of cases of pneumonia in the two groups was respectively recorded at admission and after treatment. The criteria for pneumonia are: the presence of respiratory infection symptoms such as cough, sputum, fever, and confirmation of inflammatory manifestations by lung CT.
Hemoglobin | day 1 and day 90
  The examination of hemoglobin levels will be conducted through a complete blood count (CBC) test.
Total Protein | day 1 and day 90
  The examination of Total Protein levels will be conducted through a complete blood count (CBC) test.
Albumin | day 1 and day 90
  The examination of Albumin levels will be conducted through a complete blood count (CBC) test.
Prealbumin | day 1 and day 90
  The examination of Prealbumin levels will be conducted through a complete blood count (CBC) test.
body weight | day 1 and day 90
  body weight was assessed with weight scale
upper arm circumference | day 1 and day 90
  upper arm circumference was assessed with the tape.
Penetration-Aspiration Scale | day 1 and day 90
  Penetration-Aspiration Scale is an 8-point scale that measures selected aspects of airway penetration and aspiration. The score is determined primarily by the depth to which material passes in the airway and whether material entering the airway is expelled. The scores were negative correlated with the swallowing function
Functional Oral Intake Scale for Infants | day 1 and day 90
  The Functional Oral Intake Scale for Infants was also used to assess the feeding and swallowing abilities of infants. The The Functional Oral Intake Scale for Infants provided a systematic framework for evaluating an infant's level of oral intake. The minimum values are 0 and maximum values are 7, and higher scores mean a better outcome, better swallowing ability.
Feeding amount | day 1, day 11, day 21, day 31, day 41, day 51, day 61, day 71, day 81 and day 90
  The volume of all nutrients obtained by the pediatric patients through tube feeding on the same day would be recorded, excluding water, unit: milliliter.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Study Chair — Site Coordinator of United Medical Group
Locations (1):
- Center Rehabilitation Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No